CLINICAL TRIAL: NCT00964548
Title: Dantrolene in the Treatment of Cerebral Vasospasm After Subarachnoid Hemorrhage - a Phase 1 Study
Brief Title: Safety Study of Dantrolene to Treat Cerebral Vasospasm After Subarachnoid Hemorrhage
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Susanne Muehlschlegel, Study Principle Investigator, University of Massachusetts, Worcester
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-13076
Record Dates: First submitted 2009-08-23; First posted 2009-08-25 (Estimated); Results first posted 2012-05-25 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-04

CONDITIONS: Cerebral Vasospasm After Subarachnoid Hemorrhage
Keywords: vasospasm; subarachnoid hemorrhage; neurocritical care; dantrolene; vasorelaxation
MeSH Terms: conditions — Subarachnoid Hemorrhage; Aneurysm | interventions — Dantrolene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dantrolene (low dose) (Experimental)
  Interventions: Drug: Dantrolene
- Dantrolene (high dose) (Experimental)
  Interventions: Drug: Dantrolene

INTERVENTIONS:
Drug: Dantrolene — 1.25 mg/kg IV once over 60 min
  Arms: Dantrolene (low dose)
Drug: Dantrolene — 2.5 mg/kg IV once over 60 min
  Arms: Dantrolene (high dose)

SUMMARY:
Subarachnoid hemorrhage (SAH) is a devastating acute brain injury due to bleeding onto the brain surface from a ruptured aneurysm. Cerebral vasospasm (cVSP; critical narrowing of brain arteries) is a known complication after SAH and significantly increases disability and death after SAH. Vasospasm is difficult to treat and can lead to stroke. Animal studies have shown that the muscles in the artery wall play a role in cVSP.

Dantrolene has been FDA approved and extensively used in clinical practice as a muscle relaxant for more than 30 years. It has been shown to provide some benefit in animal studies of cVSP, as well as in a small number of humans. Therefore, we plan to undertake this study to evaluate the safety and tolerability of treatment with dantrolene in patients with cVSP after SAH, and to determine the maximal tolerated dose to be used in future studies to determine if treatment with Dantrolene can improve the outcome of patients with cVSP after SAH.

DETAILED DESCRIPTION:
Our main objectives are: 1) to evaluate the safety and tolerability of varying doses of dantrolene, by determining the treatment related adverse events, in participants with cVSP after SAH; and 2) to determine the maximal tolerated dose to be adopted in subsequent studies and 3) to determine efficacy trends of dantrolene on brain vessels as assessed by ultrasound of brain vessels (transcranial Doppler).

We hypothesize that dantrolene is well-tolerated and has minimal serious adverse effects in patients with cVSP after SAH. The results can potentially bring a new treatment to patients with SAH. cVPS after SAH is a frequent cause of disability and death. A successful study demonstrating the safety of dantrolene in would be of considerable public health significance.

ELIGIBILITY:
Inclusion Criteria:

* Participants with aneurysmal SAH admitted to the Massachusetts General Hospital NeuroICU (Blake 12) and undergoing standard-of-care daily transcranial doppler (TCD).
* Participants with unilateral or bilateral anterior cerebral artery (ACA), middle cerebral artery (MCA), posterior cerebral artery (PCA), or basilar artery vasospasm as defined by the following TCD criteria
* a >50% mean velocity increase from the baseline mean TCD velocity (baseline is the first TCD measurement, usually within 24hrs of admission), or
* peak systolic TCD velocities of 200 cm/s or higher in the MCA or ACA (for MCA with a concurrent ipsilateral LR of 3.0 or higher), or peak systolic TCD velocities of 120 cm/s or higher in the PCA or basilar artery, or
* any daily 100 cm/s peak systolic TCD velocity increase from the previous day, or
* any longitudinal mean TCD velocity increase of 80 cm/s or more

Exclusion Criteria:

* Inability to obtain consent from patient or health care proxy
* Age < 18 years
* Pregnancy
* Traumatic SAH
* Known allergy to dantrolene
* Prior history of cirrhosis or hepatitis B/C, or any two of the following three liver enzymes elevated to greater than: ALT >165 Units/L, AST >120 Units/L, alkaline phosphatase >345 Units/L (three times upper limit of normal)
* Participants on verapamil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Muehlschlegel, MD, Principal Investigator — UMASS Medical School; John R Sims, MD, Study Director — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - UMASS Memorial Medical Center/UMASS Medical School, Worcester, Massachusetts

REFERENCES:
- [Background] Muehlschlegel S, Rordorf G, Bodock M, Sims JR. Dantrolene mediates vasorelaxation in cerebral vasoconstriction: a case series. Neurocrit Care. 2009;10(1):116-21. doi: 10.1007/s12028-008-9132-5. Epub 2008 Aug 12. PMID 18696267
- [Background] Salomone S, Soydan G, Moskowitz MA, Sims JR. Inhibition of cerebral vasoconstriction by dantrolene and nimodipine. Neurocrit Care. 2009;10(1):93-102. doi: 10.1007/s12028-008-9153-0. Epub 2008 Oct 16. PMID 18923817
- [Background] Muehlschlegel S, Sims JR. Dantrolene: mechanisms of neuroprotection and possible clinical applications in the neurointensive care unit. Neurocrit Care. 2009;10(1):103-15. doi: 10.1007/s12028-008-9133-4. Epub 2008 Aug 12. PMID 18696266
- [Result] Muehlschlegel S, Rordorf G, Sims J. Effects of a single dose of dantrolene in patients with cerebral vasospasm after subarachnoid hemorrhage: a prospective pilot study. Stroke. 2011 May;42(5):1301-6. doi: 10.1161/STROKEAHA.110.603159. Epub 2011 Mar 31. PMID 21454813

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates: June 2007 - October 2008 Massachusetts General Hospital NeuroICU
Pre-assignment Details: Participants were excluded from study if transcranial doppler (TCDs) did not show elevated velocities suggesting vasospasm. See inclusion criteria regarding specifics. After enrollment, TCDs were repeated. Once the repeat TCD confirmed elevated velocities suggestive of vasospasm, a single dose of IV dantrolene was infused.
Groups:
- Dantrolene (Low Dose): Single dose of Dantrolene 1.25 mg/kg infused over 60 min.
- Dantrolene (High Dose): Single dose of Dantrolene 2.5 mg/kg infused over 60 min.
Period: Overall Study
Arm/Group | Dantrolene (Low Dose) | Dantrolene (High Dose)
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dantrolene (Low Dose) | Dantrolene (High Dose) | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 42 (9) | 44 (10) | 43 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Hemodynamic Parameters (Change From Baseline Systolic Blood Pressure (Pre-infusion) Over Time Until 135 Minutes Post-infusion)
Description: Systolic Blood Pressure (Change from baseline systolic blood pressure (pre-infusion) over time until 135 minutes post-infusion).
Time Frame: baseline until 135 minutes post-infusion
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Dantrolene (Low Dose) | Dantrolene (High Dose)
Number analyzed (Participants) | 5 | 5
mmHg | -8 [-26 to 10] | -3.4 [-19 to 12]

2. Secondary Outcome: Transcranial Doppler Peak Systolic Velocity (Change From Baseline Peak Systolic Velocity (Pre-infusion) Over Time Until 135 Minutes Post-infusion)
Description: Peak Systolic Velocity of vessel in vasospasm (Change from baseline peak systolic velocity (pre-infusion) over time until 135 minutes post-infusion).
Time Frame: baseline until 135 minutes post-infusion
Measure: Mean (95% Confidence Interval); unit: cm/s
Arm/Group | Dantrolene (Low Dose) | Dantrolene (High Dose)
Number analyzed (Participants) | 5 | 5
cm/s | -30 [-47 to 12] | -26 [-56 to 8]

3. Secondary Outcome: Transcranial Doppler Mean Flow Velocity (Change From Baseline Mean Flow Velocity (Pre-infusion) Over Time Until 135 Minutes Post-infusion)
Description: Mean flow velocities of vessel in vasospasm (Change from baseline mean flow velocity (pre-infusion) over time until 135 minutes post-infusion).
Time Frame: baseline until 135 minutes post-infusion
Measure: Mean (95% Confidence Interval); unit: cm/s
Arm/Group | Dantrolene (Low Dose) | Dantrolene (High Dose)
Number analyzed (Participants) | 5 | 5
cm/s | -18 [-32 to -3] | -13 [-34 to 8]

ADVERSE EVENTS:
Time Frame: Up to 24 hours after Dantrolene infusion
Arm/Group | Dantrolene (Low Dose) | Dantrolene (High Dose)
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dantrolene (Low Dose) (N=5) | Dantrolene (High Dose) (N=5)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) — Hypotension during infusion due to vasopressor infusion stop (ran out during infusion, leading to BP drop).
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dantrolene (Low Dose) (N=5) | Dantrolene (High Dose) (N=5)
Venous Irritation (Vascular disorders) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations of this trial include the small n. No power analysis was performed, but rather a convenience sample was chosen as this was a proof-of-concept study. Transcranial Doppler measurements are operator dependent.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No